CLINICAL TRIAL: NCT07350278
Title: Comparing Virtual Reality Simulation to High Fidelity Simulation as an Educational Modality for Electroconvulsive Therapy Training: A Non-Inferiority Study
Acronym: ECT-SIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Fahad Alam, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6838
Record Dates: First submitted 2025-12-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Education, Medical, Undergraduate; Electroconvulsive Therapy; Virtual Reality Simulation
Keywords: virtual reality; mannequin; education; electroconvulsive therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled non-inferiority study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Simulator Group (Experimental): Participants randomized to this group will practice electroconvulsive therapy (ECT) administration using a virtual reality (VR) ECT simulator.
  Interventions: Other: Virtual Reality electroconvulsive therapy simulator
- Mannequin Simulator Group (Active Comparator): Participants randomized to this group will practice electroconvulsive therapy (ECT) administration using a mannequin ECT simulator.
  Interventions: Other: Mannequin Simulator

INTERVENTIONS:
Other: Virtual Reality electroconvulsive therapy simulator — A virtual reality (VR)-based simulator for electroconvulsive therapy (ECT) practice. Users will go through tutorials on how to use the VR equipment and be guided through an ECT tutorial, then they can practice ECT with no guidance at 3 distinct difficulty levels. Level 1 of the simulator will contain ECT scenarios with very few patient conditions that need additional consideration. Level 2 will contain more patient conditions that need additional consideration, as well as a chance for adverse events to occur during treatment. Level 3 will contain many patient conditions that require the user to consider when deciding how to provide ECT, as well as a high chance of adverse events occurring. Users will be shown how well they did after completing a run of a scenario.
  Arms: VR Simulator Group
Other: Mannequin Simulator — A mannequin that users can use to practice electroconvulsive therapy (ECT) administration on. Users will be provided a mannequin and ECT equipment, as well as a scenario check-list to go through.
  Arms: Mannequin Simulator Group

SUMMARY:
The goal of this prospective, open-label non-inferiority randomized controlled trial is to investigate if Virtual Reality (VR) based simulation are an effective training tool for novice medical trainees. The main questions it aims to answer are:

* Is the VR-based electroconvulsive therapy (ECT) training program non-inferior to traditional, mannequin-based ECT training programs in fostering ECT skill acquisition?
* What are the changes in confidence in administering ECT, as well as number of training repetitions completed in the VR and mannequin training groups?
* What is the ease of use of the VR-based ECT training program? Researchers will compare the VR-based ECT training program to a mannequin-based ECT training program to see if the VR-based ECT training program is comparable to traditional methods at training for ECT.

Participants will:

* Complete an ECT skills assessment at the beginning and end of the study session.
* Watch a 30-minute didactic ECT lecture video.
* Be randomized to either the VR ECT simulation group or the mannequin ECT simulation group and be given 30 minutes to practice ECT administration with their assigned education tool.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is one of the most validated treatments for major depressive disorder (MDD), particularly treatment-resistant MDD where patients do not respond to at least two full courses of antidepressant medications and one full course of cognitive behavioral therapy. Despite its proven efficacy and safety, ECT is still heavily underutilized compared to other treatments. One of the causes for ECT underutilization is a stagnation in the growth in numbers of ECT-competent practitioners over the past 30 years. This issue stems from a lack of formal, standardized, and effective ECT training for medical trainees.

Virtual reality (VR) technology has been emerging as a promising medium for medical training due to its ability to create highly immersive and interactive simulations. Compared to traditional simulation mediums such as high-fidelity mannequins, VR is advantageous in that the cost of repeated use is low, usage of VR is not limited to a specialized facility, and VR training programs can be easily disseminated. VR-based simulations for medical training has already been developed for disciplines such as anesthesiology, where VR-based simulation tools are used to aid the learning of techniques such as bronchoscopy. However, there currently lacks a validated VR training tool for ECT.

Here the investigators propose to study a VR-based ECT training simulation, and see if it is non-inferior to a mannequin-based ECT training simulation. The mannequin-based simulation represents experiential learning, which is one of the ways ECT is currently taught.

Medical students who have not received any ECT training (N = 78) will begin the study by completing an ECT skills assessment test, where they must go through an ECT scenario on a mannequin. Afterwards, participants will watch a 30-minute didactic ECT lecture video. Participants will then be randomized to either the intervention group (VR simulation training group, N = 39) or the active control (mannequin simulation training group, N = 39). Participants will be instructed on how to use their assigned education modality, then given around 30 minutes to practice with their education modality. After the training sessions, participants will complete the ECT skills assessment test again.

The ECT skills assessment tests will be recorded, and two blinded raters will rate the ECT competency of the participant based on an ECT competency scale. Participants will also be asked how confident they are at administering ECT before and after the training sessions, as well as how many training repetitions they completed during their session.

ELIGIBILITY:
Inclusion Criteria:

* Is a medical student at the University of Toronto
* Has not received formal ECT training before

Exclusion Criteria:

* Visual or hearing impairment that does not allow the participant to use VR.
* History of significant motion sickness.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Electroconvulsive Therapy Objective Structured Assessment of Technical Skills (ECT-OSATS) | Before and after the study educational intervention administration (day 1)
  A comprehensive ECT proficiency assessment tool including a technical skills checklist and a global performance rating scale. The technical skills checklist includes specific tasks during ECT administration that need to be completed to ensure a successful ECT delivery. Scores for each task can range from 1 - "Not Done" to 3 - "Done Correctly". Higher scores indicate better performance. The global performance rating scale includes items such as "Efficiency", "Knowledge", "Communication", and "Overall Impression of Performance" of the participant's ECT administration session as a whole. Scores can range from 1 - 5, with higher scores indicating a more positive outcome. The rating scale culminates with a "Global Impression of Pass or Fail", with options of "Fail" - the participant cannot perform ECT independently, or "Pass" - the participant can perform ECT independently. The ECT-OSATS was adapted from Rabheru et al. (2013).

SECONDARY OUTCOMES:
VR System Usability Scale (SUS) | After the study educational intervention administration (day 1)
  A questionnaire asking about the user's experience in their use of virtual reality technology. It is a 8-item questionnaire rated on a 5-point Likert scale with options of "Strongly Agree", "Somewhat Agree", "Neutral", "Somewhat Disagree", and "Strongly Disagree". Each choice is also associated with a numbered score, from "Strongly Agree" at 1 to "Strongly Disagree" at 5. Depending on the question, higher scores could indicate a more positive or a more negative outcome. E.g., for the question "I thought the VR system was easy to use", a higher score would indicate a more negative outcome. Conversely, for the question "I found the VR system unnecessarily complex", a higher score would indicate a more positive outcome. Scores will be adjusted depending on if the question rates higher scores as a positive or negative outcome. Adjusted scores will be summed, then multiplied by 2.5 and divided by 80 to yield a final system usability score out of 100. Adapted from Brooke, John (1995).
Rate of Learning Questionnaire | Before and after the study educational intervention administration (day 1)
  A 3-item questionnaire examining the participant's confidence in performing ECT at baseline and at end of study, as well as the number of practice repetitions the participant completed during the education intervention session. Confidence in performing ECT is assessed on a 3-point scale ranging from "Not At All" to "Very confident", with "Very Confident" being a more positive outcome. Practice repetitions are defined as the number of times the participant completed ECT training scenarios during their education intervention session.

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Dr. Alam, MD, FRCPC, MHSc, Principal Investigator — Sunnybrook Research Institute; Peter Giacobbe, MD, MSc, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be made available upon reasonable request to study PI following publication of full trial results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No interim analysis plan is in place, so data will be available following publication of the primary results after trial completion.
Access Criteria: Data and supporting information will be made available following reasonable request directly to study PI.